CLINICAL TRIAL: NCT00850291
Title: Prospective, Controlled, Randomized Study of Economisation of the Preparation in Partial Duodenopancreatectomy Using an Electrosurgical Sealing Device Versus Traditional Methods
Brief Title: Economisation of Whipple Resection Using Electrosurgical Sealing Device
Acronym: SEAL
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: 2907
Record Dates: First submitted 2009-02-23; First posted 2009-02-24 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Duodenopancreatectomy
Keywords: Partial duodenopancreatectomy using electrosurgical vessel sealing device

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Electrosurgical vessel sealing device
- 2: traditional surgical methods:stitches and ligations

SUMMARY:
Including 89 randomised patient, the studies aim is to determine whether an economisation and/or improvement in terms of operating time, drainage fluid, blood loss, time of hospitalisation can be found using an electrosurgical sealing device versus traditional surgical methods such as stitches an ligations.The study is performed for patients undergoing partial pancreatoduodenectomy.

ELIGIBILITY:
Inclusion Criteria:

* resectable tumor

Exclusion Criteria:

* palliative resection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients planned for partial pancreatoduodenectomy for pancreatic head carcinoma, periampullary carcinoma, chronic pancreatitis and other benign lesions.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2008-05; Primary Completion 2010-02 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob R. Izbicki, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- UH Eppendorf, Hamburg, Germany

REFERENCES:
- [Background] Ujiki MB, Talamonti MS. Guidelines for the surgical management of pancreatic adenocarcinoma. Semin Oncol. 2007 Aug;34(4):311-20. doi: 10.1053/j.seminoncol.2007.05.004. PMID 17674959
- [Derived] Uzunoglu FG, Bockhorn M, Fink JA, Reeh M, Vettorazzi E, Gawad KA, Bogoevski D, Vashist YK, Tsui TY, Koenig A, Mann O, Izbicki JR. LigaSure vs. conventional dissection techniques in pancreatic surgery--a prospective randomised single-centre trial. J Gastrointest Surg. 2013 Mar;17(3):494-500. doi: 10.1007/s11605-012-2107-z. Epub 2012 Dec 19. PMID 23250820